CLINICAL TRIAL: NCT03487575
Title: Integrated Electronic and Care Manager Support Intervention For Caregivers of Adolescents With Suicidal Behavior--Open Trial
Brief Title: Integrated Intervention for Caregivers--Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Duke University (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00055566-OT
Record Dates: First submitted 2018-03-16; First posted 2018-04-04 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Distress; Maternal; Self-Efficacy; Parenting; Suicide
Keywords: Adolescent; Parental Support; Parental Coping
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open trial (Experimental)
  Interventions: Behavioral: Open trial

INTERVENTIONS:
Behavioral: Open trial — Integrated electronic support and care support manager contact

SUMMARY:
Adolescents who have been hospitalized for suicidal behavior are at risk for engaging in additional suicidal behavior. After hospitalization, parents or guardians are typically asked to be responsible for helping to prevent further suicidal behavior. This can include monitoring the youth, making sure the home is safe, getting the youth any needed treatment, and balancing the parents' expectations of the youth with the understanding that the youth is in a vulnerable state. Even with these efforts by parents, adolescents often have additional crisis situations. The goal of this study is to develop and test an integrated electronic and care support service intervention for parents of suicidal youth. It is expected that this intervention will help parents/guardians in the roles of caring for suicidal youth after discharge from the hospital. This open trial will assess the feasibility of this intervention for a separate pilot randomized controlled trial to compare the intervention to enhanced treatment as usual.

DETAILED DESCRIPTION:
Adolescents who have been hospitalized for suicidal behavior are at high risk for engaging in additional suicidal behavior. Following hospitalization, parents or guardians are typically tasked with helping to prevent further suicidal episodes by monitoring youth, ensuring safety in the home, helping youth receive needed care, and parenting in a way that balances expectations for appropriate behavior with recognition of the vulnerable status of the adolescents. Despite parental efforts, adolescents often have additional crises, which sometimes culminate in emergency department visits and repeat hospitalizations. Findings from the principal investigators' recent longitudinal study of mothers after adolescent hospitalization for suicide attempts (Impact of Adolescent Hospitalization on Parents) suggested that the period of time following discharge from the hospital can be a very important time for providing services and supports to youth and families. Parents in that study described emotional distress (e.g., depression, anxiety) and reduced parenting self-efficacy, and indicated a need for more information about suicidal youth and the treatment needs of these youth, parenting and monitoring of suicidal youth, and support in navigating the treatment system.

Given these needs, the purpose of this study is to develop, refine, and preliminarily test an integrated electronic and care support service intervention for caregivers of adolescents who have recently engaged in suicidal behavior. It is expected that such an intervention will provide needed information and supports to parents, increase parenting self-efficacy, increase parents' ability to follow safety plans in the home, reduce parents' emotional distress, and help parents access needed services in the community. As a consequence of these proximal outcomes, it is expected that the intervention will help facilitate treatment engagement and follow through for youth and caregiver, and reduce use of emergency mental health services and hospitalizations.

In the context of an open trial, the primary aim is to assess the feasibility of this intervention, and to use experiences from implementing the intervention and feedback from caregivers and care support managers to refine the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Biological, adoptive, or step-parent (step-parent defined as by marriage or live-in partner of at least 5 years) of an adolescent. If an adolescent has more than one parent, parents will be asked to designate the primary contact or participant for this study (only one parent for an adolescent may participate).
* The adolescent is 13-19 years of age
* The adolescent was psychiatrically hospitalized due to any range of suicidal behaviors (i.e., suicide attempt, interrupted suicide attempt, aborted suicide attempt) in the last two weeks
* The parent lives with the adolescent
* The parent has a cell phone and is capable of texting (i.e., has knowledge of how to text and has a data plan that allows for texting)

Exclusion Criteria:

* Parents whose primary language is not English and are unable to read or speak English, as all materials will be initially developed in English only
* Parents who have a reported intellectual disability (per inpatient staff)
* Parents whose adolescent is not discharged directly home (e.g., adolescent is sent to a group home, residential treatment facility, or home of a relative following hospitalization)
* Adolescents who have an intellectual disability (per inpatient staff or as reflected by current school placement) or have active psychosis, as the needs of both parent and youth may be different than those without an intellectual disability or active psychosis and are not specifically addressed in the proposed developing intervention

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Change in parental distress as assessed with SCL-90-R | Baseline (hospitalization), and at 3- and 6- months following discharge
  To assess severity of depression, anxiety, and hostility, parents will be administered the Symptom Checklist - 90 (SCL-90-R). The SCL-90-R yields scores along several dimensions: Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. The scale range for each dimension is a T-score of 0-100, with higher scores representing greater problem severity.
Change in parental self-efficacy as assessed with PSOC | Baseline (hospitalization), and at 3- and 6- months following discharge
  Facets of parental self-efficacy will be assessed with the Parenting Sense of Competence Scale (PSOC), which measures sense of self-efficacy and satisfaction with parenting. It has a scale range of 17-102, with higher scores indicating a greater parenting sense of competency. It has been used with parents of children and adolescents.
Change in parental self-efficacy as assessed with "Me as a Parent" Parent Self-Regulation scale | Baseline (hospitalization), and at 3- and 6- months following discharge
  Facets of parental self-efficacy will be assessed with the "Me as a Parent" Parenting Self-Regulation scale, which assesses constructs such as sense of effectiveness, sense of control as a parent, ability to manage situations with children (a central concept for the current study), and parental self-management (planful parenting activities). The scale range is 16 - 80, with higher scores representing a greater parental sense of self-regulation. It has been used with parents of children and adolescents.
Change in parenting practices as assessed with Alabama Parenting Practices Questionnaire | Baseline (hospitalization), and at 3- and 6- months following discharge
  The Alabama Parenting Practices Questionnaire will be used to assess parenting behaviors. For purposes of our study, investigators will focus on the parental involvement subscale (10 items), the positive parenting subscale (6 items), the monitoring and supervision subscale (10 items), and the inconsistent discipline scale (6 items). The scale ranges are 10-50 for the 10-item subscales, and 6-30 for the 6-item subscales. Higher scores denote better outcomes for the parental involvement and positive parenting subscales, whereas higher scores denote worse outcomes for the monitoring/supervision and inconsistent discipline subscales.
Change in parent reports of adolescent suicidal behavior as assessed with C-SSRS | Baseline (hospitalization), and at 3- and 6- months following discharge
  Parental reports of adolescent suicidal ideation and behaviors following hospitalization will be assessed with selected queries from the Columbia - Suicide Severity Rating Scale (C-SSRS). This measure does not have an overall scoring range, but it does include a suicidal ideation intensity rating with a range 0-25. In general, a greater number of endorsed items and/or a higher suicidal ideation intensity rating denote greater suicidal risk.
Change in child emotional and behavioral problems as assessed with CBCL | Baseline (hospitalization), and at 3- and 6- months following discharge
  To provide some contextual information at each assessment, parents at baseline hospitalization only will complete the Achenbach Child Behavior Checklist (CBCL). The CBCL is a widely used parent-report scale. The measure includes 20 subscales, each having a T-score range of 50-100, with higher scores denoting greater psychological and behavioral problems.

SECONDARY OUTCOMES:
Change in parent perceptions of support and safety monitoring as assessed with a series of likert rating questions | Through study completion, up to 6 months following discharge
  Using a series of likert rating questions, investigators also will assess the degree to which parents feel provided with information regarding their child's condition and the management of their child in the home, and the degree to which parents feel supported by the intervention and by mental health professionals. Investigators will use likert scales at formal assessment points to assess perceived success and confidence in monitoring youth and following safety plans in the first month after hospitalization, and during any other times of high risk. In addition to formal assessments, the care support manager will use ratings during regular check-ins to gauge the degree to which parents' needs are being met.
Adolescent service use assessed with CASA and treatment records | Baseline (hospitalization), and at 3- and 6- months following discharge
  The semi-structured interview-based Child and Adolescent Services Assessment-Parent Interview-Version 5.0 (CASA) will be used to assess emergency department visits and repeat hospitalizations; duration and frequency of adolescent involvement with specialty mental health services (therapists, psychiatrists, etc.) following hospitalization; and attitudes about service use for adolescents. In addition, with consent/assent of parents and adolescents, investigators will obtain adolescents' treatment records to verify contacts with mental health providers. This measure does not have an overall scale range.
Cost information assessed with measure of time spent | Up to 6 months following discharge
  Time spent by the care support manager in patient contacts, preparation, and documentation will be tracked to estimate potential costs. These data will be preliminary due to the early phase of intervention development, but will set the stage for scalability efforts and later well-powered cost-effectiveness studies.
Assessment of the patient satisfaction and acceptability of the intervention assessed with Client Satisfaction Questionnaire | Through study completion, up to 6 months following discharge
  To assess patient satisfaction and acceptability of the intervention, investigators will administer the Client Satisfaction Questionnaire. This measure has a range of 8-32, with higher scores indicating greater satisfaction. Following Mohr et al. (2011), additional indices of the acceptability and usability of the intervention will include the degree to which parents use the mHealth application over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie S Daniel, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
In order to adhere to the goal of data sharing among researchers, investigators will share data from this study via the National Database for Clinical Trials related to Mental Illness (NDCT). Based on the procedures outlined on the NDCT web site, investigators will collect information necessary to generate a Global Unique Identifier (GUID), a universal subject identifier, for each participant. No personal identifying information, nor data that could be used deductively to identify participants, however, will be shared with other researchers, particularly given the relatively small size of the data set. The GUID will allow sharing of information across research studies. Research participants will be informed of the Resource Sharing Plan in the consent forms for participation in the studies, using text similar to the example plain language text for informed consent forms provided by the NDCT.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Investigators will begin uploading raw data to the NDCT system semiannually (January 15, July 15) after data collection has begun. All data will be shared prior to the end of the grant.
Access Criteria: Data will be shared with researchers who have access to the National Database for Clinical Trials related to Mental Illness (NDCT).

DOCUMENTS (1):
  • Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03487575/ICF_000.pdf